CLINICAL TRIAL: NCT06011954
Title: Use-result Surveillance for PADCEV Injection 20 mg and 30 mg (Enfortumab Vedotin) in South Korea
Brief Title: A Study to Survey Adults in South Korea With Cancer Who Receive PADCEV Injection
Status: Recruiting | Type: Observational
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 7465-PV-0001
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Urothelial Cancer
Keywords: Urothelial Cancer; Bladder Cancer; enfortumab vedotin; PADCEV
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PADCEV: Patients who receive PADCEV Injection 20 mg and 30 mg (enfortumab vedotin) in routine clinical practice according to the drug label approved at the time of marketing authorization.
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Enfortumab Vedotin — Intravenous
  Other Names: PADCEV; ASG-22CE

SUMMARY:
Enfortumab vedotin (or PADCEV Injection) is a treatment for cancer in the bladder lining (urothelial cancer). PADCEV Injection is now available to treat this cancer.

People in this study will be adults in South Korea with locally advanced or metastatic urothelial cancer. Metastatic means the cancer has spread to other parts of the body. During their care, the person's doctor will have prescribed PADCEV Injection and other medicines to treat their cancer. People in the study will be treated according to their clinic's standard practice. This study is about collecting information only.

This study will survey people who know they are receiving PADCEV Injection. The aims of the study are to check outcomes of treatment with PADCEV and record any medical problems during the study.

Once a doctor has prescribed PADCEV Injection, a person in the study will be observed for up to 48 weeks (about 1 year) after their first dose. During this time, a person's medical records will be reviewed to check for any medical problems and to follow the condition of their cancer. If a person in the study stops taking PADCEV Injection sooner than 48 weeks, records will be reviewed until 30 days (1 month) after each person's last dose of PADCEV Injection or until they start a different medicine for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive treatment with PADCEV Injection, according to the approved local label.

Exclusion Criteria:

* Patients with any contraindication for PADCEV Injection, according to the approved local label.
* Patients who receive or are going to receive any investigational medicine during the observation period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Adult participants with locally advanced (LA) or metastatic urothelial cancer (mUC) in South Korea who are prescribed PADCEV Injection and have previously received a Programmed death receptor-1 or Programmed death-ligand 1 inhibitor and have received a platinum containing chemotherapy.
  * Adult participants with LA or mUC in South Korea who are prescribed PADCEV Injection in combination with pembrolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an Adverse Event | Up to 48 weeks after the first administration of PADCEV
  Adverse events (AEs) will be summarized using MedDRA. An AE is defined as any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Number of patients with an adverse drug reaction (ADR) | Up to 48 weeks after the first administration of PADCEV
  An ADR is defined as any noxious and unintended response associated with the use of a drug in humans, at any dose, where a causal relationship is at least a reasonable possibility.
Number of patients with a serious AE (SAE) | Up to 48 weeks after the first administration of PADCEV
  An AE is considered "serious" if it results in death or is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is a medically important event or reaction.
Number of patients with a serious ADR (SADR) | Up to 48 weeks after the first administration of PADCEV
  An ADR is considered "serious" if it results in death or is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is a medically important event or reaction.
Number of patients with an unexpected AE (UAE) | Up to 48 weeks after the first administration of PADCEV
  An UAE is an AE that the nature or severity of which is not consistent with the information in the approved Korean label.
Number of patients with an unexpected ADR (UADR) | Up to 48 weeks after the first administration of PADCEV
  An UADR is defined as an unexpected adverse drug reaction.
Number of patients with an important risk | Up to 48 weeks after the first administration of PADCEV
  An important risk is classified as an important identified risk and an important potential risk.
  An identified risk is defined as the risk that correspond to undesirable clinical outcomes, with sufficient scientific evidence that the undesirable clinical outcome is caused by the drug."Important Identified Risks" are identified risks that have the potential to affect the risk-benefit balance of a product.
  An potential risk is defined as the risk that correspond to undesirable clinical outcomes, with some, but not sufficient, evidence to estimate that the undesirable clinical outcome is caused by the drug."Important Potential Risks" are potential risks that have the potential to affect the risk-benefit balance of a product.

SECONDARY OUTCOMES:
Overall survival | Up to 48 weeks after the first administration of PADCEV
  Overall survival (OS) is defined as time from start of PADCEV to death.
Progression free survival | Up to 48 weeks after the first administration of PADCEV
  Progression free survival (PFS) is defined as time from start of PADCEV to progressive disease (PD) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Korea, Inc.
Locations (18):
- South Korea (18):
  - Site KR82001, Goyang-si, Gyeonggi-do
  - Site KR82012, Suwon, Gyeonggi-do
  - Site KR82008, Suwon, Gyeonggi-do
  - Site KR82007, Jeollanam-do, Jeollanam-do
  - Site KR82013, Jeonju, Jeonbuk-do
  - Site KR82015, Busan
  - Site KR82010, Busan
  - Site KR82009, Busan
  - Site KR82016, Busan
  - Site KR82014, Daegu
  - Site KR82018, Daejeon
  - Site KR82004, Incheon
  - Site KR82002, Seoul
  - Site KR82005, Seoul
  - Site KR82003, Seoul
  - Site KR82017, Seoul
  - Site KR82006, Seoul
  - Site KR82011, Seoul

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.